CLINICAL TRIAL: NCT01354626
Title: Influence of Increasing Dietary Protein on Hepatic Fat Accumulation and Postprandial Metabolism
Brief Title: Dietary Protein and Hepatic Fat Accumulation
Acronym: LiF-Pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LiF-Pro
Record Dates: First submitted 2011-05-13; First posted 2011-05-17 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Hepatic Fat Accumulation; Nonalcoholic Fatty Liver Disease
Keywords: Hepatic fat accumulation; Dietary protein; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Dietary Proteins; Diet; Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat diets (Experimental): High-fat-Low-protein or High-fat-high-protein
  Interventions: Other: dietary protein
- Control group (Other): Low-protein-low-fat (according to healthy eating guidelines)
  Interventions: Other: low-protein

INTERVENTIONS:
Other: dietary protein — in the low-protein group 13EN% of protein will be provided in the diet; in the high-protein 25EN% of protein will be provided
  Other Names: diet
  Arms: High fat diets
Other: low-protein — The control group will get a diet which is according to healthy eating guidelines.
  Other Names: diet
  Arms: Control group

SUMMARY:
The objective of this study is to investigate the potential beneficial effect of increasing protein in the diet in order to decrease hepatic lipid accumulation on a high-fat diet.

The investigators hypothesize that increasing protein in a high-fat diet suppresses lipid accumulation in the liver, and that changes in (hepatic) fat handling underlie this reduced lipid accumulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* body mass index (BMI) 18-25 kg/ m2;
* stable dietary habits;
* physical activity levels.
* caucasian

Exclusion Criteria:

* Unable or unwilling to comply with study procedures;
* not caucasian
* Unstable body weight (weight gain or loss > 3 kg in the past three months);
* Moderate intense physical activity (exercise) for more than 4 hours/week;
* (Chronic) disease which might influence the study outcomes e.g. diabetes mellitus or any other endocrine disorder, active cardiovascular disease, hepatic disease, renal disease, cancer;
* Family history of diabetes mellitus;
* Use of medication, except incidental use of paracetamol;
* Abuse of drugs;
* Alcohol consumption of more than 14 glasses per week;
* Participation in another biomedical study within 1 months prior to the first screening visit;
* Contraindications to MRI scanning. These contraindications include patients with one of the following conditions:
* Claustrophobia;
* Central nervous system aneurysm clips;
* Implanted neural stimulator;
* Implanted cardiac pacemaker or defibrillator;
* Cochlear implant;
* Ocular foreign body (e.g. metal shavings);
* Insulin pump;
* Metal shrapnel or bullet;
* Or metal containing corpora aliena in the eye of brains.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
hepatic fat accumulation | baseline, 2 weeks, 4 weeks

SECONDARY OUTCOMES:
Biomarkers of liver function/hepatic steatosis | baseline, 2 weeks, 4 weeks
  Biomarkers of liver function/hepatic steatosis: ALT, AST, C-reactive protein
Circulating cytokines | baseline, 2 weeks, 4 weeks
  adiponectin, TNF-α
Postprandial lipid metabolism | 2 weeks, 4 weeks
  Postprandial lipid metabolism will be assessed by means of a meal challenge with the use of stable isotope tracer
Glucose homeostasis | baseline, 2 weeks, 4 weeks
  Glucose homeostasis will be assessed with the homeostatic model assessment (HOMA) index in fasting blood samples. In addition dynamic indexes will be determined from the meal challenge.
Adipose tissue gene expression | 2 weeks, 4 weeks
Peripheral blood mononuclear cells gene expression (PBMC's). | baseline, 2 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Rietman A, Schwarz J, Blokker BA, Siebelink E, Kok FJ, Afman LA, Tome D, Mensink M. Increasing protein intake modulates lipid metabolism in healthy young men and women consuming a high-fat hypercaloric diet. J Nutr. 2014 Aug;144(8):1174-80. doi: 10.3945/jn.114.191072. Epub 2014 Jun 4. PMID 24899158